CLINICAL TRIAL: NCT04738643
Title: Improving Tobacco Treatment Rates for Cancer Patients Who Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 04019; SAP#4100083101 (Other Grant/Funding Number: Commonwealth of Pennsylvania); 832404 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Tobacco Use; Smoking; Nicotine Dependence
Keywords: Cancer; Smoking; Tobacco Use; Nicotine Dependence; Tobacco Use Treatment Service
MeSH Terms: conditions — Neoplasms; Tobacco Use; Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): TUT Service Only
- Tobacco Use Treatment Service + Varenicline Management (Experimental): TUTS + Varenicline Management
  Interventions: Other: Tobacco Use Treatment Service and Varenicline Management

INTERVENTIONS:
Other: Tobacco Use Treatment Service and Varenicline Management — The VM intervention builds upon the established TUT Service process. In addition to connecting the patient to TUT Service via electronic referral, it activates a medication management protocol that: 1) actively confirms no evidence of renal failure or pregnancy with oncology provider, 2) automates a referral to prescribing providers within the TUT Service team, prompting a call-back to patient within 24 hours, 3) provides written AVS instructions to contact TUT Service for initiation instructions and clinic appointment, and 4) pends a varenicline prescription to the medication list, ready for reconciliation by TUT Service prescribing clinicians. The protocol formalizes standard management principles for varenicline, including follow-up evaluation, pre-quit period duration, and side effect amelioration.
  Other Names: TUTS + VM; TUT Service + VM
  Arms: Tobacco Use Treatment Service + Varenicline Management

SUMMARY:
The research objective is to identify a simple, pragmatic, innovative way of enhancing Tobacco Use Treatment (TUT) rates within oncology. To investigate this possibility, the investigators propose methods that will allow them to: 1) evaluate the impact of standing orders to initiate a varenicline management protocol within outpatient cancer treatment workflow, 2) assess the potential for an EHR-based intervention to affect patient TUT behaviors, and 3) identify important facilitators and barriers that impact effectiveness of the intervention.

The investigators will assess whether including a standing order for prescription and management of varenicline (TUT Service+VM) within the workflow for cancer patients identified as current smokers will significantly increase TUT engagement rates compared to current standard of care (TUT Service alone). The investigators hypothesize that observed treatment engagement rates will be higher among clinicians exposed to TUT Service+VM than observed in clinicians exposed to TUT Service alone.

DETAILED DESCRIPTION:
To reduce all-cause and cancer-specific mortality, the 2014 Surgeon General's Report emphasized the importance of effective tobacco use treatment (TUT) in cancer care. Unfortunately, up to 50% of cancer patients who smoke prior to their diagnosis continue to do so after diagnosis and treatment. This observation has lead the National Comprehensive Cancer Network, the American Society of Clinical Oncology, and the American Association for Cancer Research to call for implementation strategies integrating TUT directly within oncology care. At this time, many cancer centers and oncology practices fall short of providing consistent, high-quality TUT; only half of cancer centers report that they identify tobacco use among patients, and very few use systematic mechanisms to encourage TUT services.

In response, the National Cancer Institute (NCI) funded the Cancer Center Cessation Initiative (C3I) in 2017 with support from the NCI Cancer Moonshot Program. C3I's aim is to help build and sustain TUT infrastructure across the nation's cancer centers, ensuring that cancer patients are systematically screened for tobacco use and provided with evidence-based smoking cessation treatment. Abramson Cancer Center's work implementing the C3I tobacco use treatment service (TUT Service) has significantly improved rates of TUT within oncology practice, however the investigators have identified a number of important social-motivational obstacles to reaching the target of universal TUT. For instance, it is known that simple changes to treatment choice architecture in the electronic health record (EHR), i.e. utilizing an "opt-out" rather than "opt-in" structure, increases TUT Service engagement in a manner similar to other contexts of cancer care. Unfortunately, there remains unacceptable variation in clinician engagement rates. One significant reason for this variation is the individual clinician's perceptions of treatment effectiveness.( A strategy used elsewhere involved utilizing opt-out orders aimed at maximizing the use of varenicline, i.e. "Varenicline Management" (VM). VM resulted in increased clinician utilization and patient cessation within a relatively controlled environment of hospital-based cardiac and pulmonary care. However, it is unknown whether this type of intervention is generalizable to the complex, challenging environment of outpatient oncology.

The goal of this study is to determine if the default for a varenicline order increases clinician referral to TUTS and/or the treatment of tobacco use. At this point, many clinicians are turning the referral order off and patients are not receiving treatment for tobacco use. A default to prescribe treatment may help override barriers to both.

Insights gained from this project form the basis of subsequent clinical trials assessing efficacy of novel implementation approaches improving uptake of evidence-based tobacco use treatment. This study is significant because the model for promoting physician behavior change is simple and pragmatic, yet has the potential to significantly impact cancer patient survival and morbidity. The study builds on previous observations made through NCI and C.U.R.E. investments, expanding the understanding of novel pharmacologic approaches to tobacco cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Currently in active practice within Medical and Radiation Oncology divisions of ACC,
2. Prescribing authority in Pennsylvania (i.e. physician, nurse practitioner, physician assistant),
3. Nonsmoker,
4. Has cared for at least one patient with tobacco use disorder in the 30 days prior to recruitment,
5. English speaking, and
6. Willing to provide informed consent to participate.

Exclusion Criteria:

1. Unwillingness to prescribe varenicline, or
2. Unwillingness to assign varenicline management to TUT Service providers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnoll R, Blumenthal D, Wileyto EP, Bauer AM, Evers-Casey S, Stevens N, Fisher T, Ware S, Jenssen BP, Wollack C, Schwartz S, Leone FT. Pilot Trial of a Behavioral Economics-Informed Clinical Decision Support Alert to Improve Inpatient Tobacco Use Treatment Rates. Nicotine Tob Res. 2025 Nov 23;27(12):2265-2272. doi: 10.1093/ntr/ntaf129. PMID 40570180

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 635 patients accrued to the study, and the 50 clinicians who saw these patients received either the intervention alert or the usual care alert depending on the arm to which they were randomized. In total, this resulted in 685 individuals who were involved in the trial.
Period: Overall Study
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Started | 425 (397 patients; 28 clinicians) | 260 (238 patients; 22 clinicians)
Patients Who Received Any Tobacco Use Treatment | 113 | 60
Completed | 425 | 260
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline information was only collected for the 635 patients who accrued to the trial, not for the 50 clinicians.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management | Total
Number analyzed (Participants) | 397 | 238 | 635
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.66 (13.73) | 57.99 (14.02) | 56.53 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 97 | 272
  Male | 222 | 141 | 363
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 383 | 231 | 614
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 294 | 181 | 475
  White | 82 | 43 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 11 | 28
Region of Enrollment [Number; unit: participants]
  United States | 397 | 238 | 635

OUTCOME MEASURES:

1. Primary Outcome: Intervention Ordering Rate
Description: Defined as the number of patients for whom any inpatient tobacco use treatment order is signed by a participating clinician, divided by the total number of patients in each arm for whom an order was pended and the alert fired
Time Frame: Up to 30 days after Initial Visit
Population: Outcome measures were only assessed for patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 397 | 238
Participants | 113 | 60

2. Secondary Outcome: Inpatient Medication Ordering Rate
Description: Defined as the number of patients for whom any inpatient tobacco use treatment medication was ordered, divided by the total number of patients in each arm for whom an order was pended and the alert fired
Time Frame: Up to 30 days after Initial Visit
Population: Outcomes were only assessed for patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 397 | 238
Participants | 73 | 41

3. Secondary Outcome: Outpatient/Discharge Medication Ordering Rate
Description: Defined as the number of patients for whom any tobacco use treatment medication was ordered upon patient discharge from the hospital, divided by the total number of patients in each arm for whom an order was pended and the alert fired
Time Frame: Up to 30 days after Initial Visit
Population: Outcomes were only assessed for patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 397 | 238
Participants | 26 | 17

4. Secondary Outcome: TUTS Referral Rate
Description: Defined as the number of inpatients for whom a referral to the health system's Smoking Cessation Program was placed, divided by the total number of patients in each arm for whom an order was pended and the alert fired
Time Frame: Up to 30 days after Initial Visit
Population: Outcomes were only assessed for patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 397 | 238
Participants | 13 | 20

5. Secondary Outcome: Quit Line Rate
Description: Defined as the total number of patients who present for quit line counseling (i.e. telephone or electronic), divided by the total number of patients referred to the Smoking Cessation Program
Time Frame: 30 Day Follow-up Assessment
Population: This outcome was only assessed for patients who were referred to the Smoking Cessation Program.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 10 | 23
Participants | 5 | 5

6. Secondary Outcome: Medication Recommendation Rate
Description: Defined as the number of patients who are recommended to receive a tobacco use treatment medication by the TUT Service staff in quit line counseling, divided by the total number of patients who present for quit line counseling
Time Frame: 30 Day Follow-up Assessment
Population: This outcome was only assessed for patients who were referred to the Smoking Cessation Program and appeared for a consult.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 5 | 5
Participants | 4 | 4

7. Secondary Outcome: Follow-up Recommendation Rate
Description: Defined as the number of patients who are recommended to receive a tobacco use treatment medication or a follow-up appointment by the TUT Service staff in quit line counseling, divided by the total number of patients who present for quit line counseling
Time Frame: 30 Day Follow-up Assessment
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
Number analyzed (Participants) | 5 | 5
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Duration of patient's stay, which averaged as approximately 11 days
Arm/Group | Usual Care | Tobacco Use Treatment Service + Varenicline Management
All-Cause Mortality (participants affected / at risk) | 0/397 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/397 | 0/238
Other Adverse Events (participants affected / at risk) | 0/397 | 0/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT04738643/Prot_SAP_000.pdf